CLINICAL TRIAL: NCT02323087
Title: Reducing Antibiotic Resistance: Improved Diagnostics and Treatment for Uncomplicated Urinary Tract Infection in General Practice, Denmark
Brief Title: Point of Care Susceptibility Testing in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anne Holm, MD PhD-student, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UCCAREWP4FLEX
Record Dates: First submitted 2014-12-11; First posted 2014-12-23 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Urinary Tract Infections
Keywords: Antibiotic resistance; Point of care tests; Primary Health Care
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Culture and susceptibility testing (Active Comparator): Urine culture and sensitivity testing will be performed using the FLEXICULT™ SSI-Urinary Kit
  Interventions: Device: FLEXICULT™ SSI-Urinary Kit
- Culture (Active Comparator): Point of care culture will be performed using ID FlexicultTM
  Interventions: Device: ID FlexicultTM

INTERVENTIONS:
Device: FLEXICULT™ SSI-Urinary Kit — Urine culture and sensitivity testing will be performed on the intervention group by means of a POCT, the FLEXICULT™ SSI-Urinary Kit. The kit is designed as an ordinary Petri dish but with higher sides. The Petri dish is divided into 6 compartments: 1 large one for quantitative analysis and 5 smaller ones for susceptibility testing (Fig. 1). The agar in each of the smaller compartments contains 1 of 5 antimicrobials: trimethoprim, sulfamethoxazole, ampicillin, nitrofurantoin and mecillinam. The agar plate is flooded with the urine specimen for a couple of seconds and then incubated at 35°C over night. The following day the plate is read. When reading the compartment for quantitative analysis the lower limit is:103 colony-forming units (cfu) per milliliter.
  Arms: Culture and susceptibility testing
Device: ID FlexicultTM — Point of care culture will be performed using ID FlexicultTM,which is a chromogenic agar plate for identification and quantitation of urinary tract pathogens. The agar plate is for cultivation of urine, which makes it possible to identify the bacteria and quantitate the amount of bacteria. Based on bacterial colony color and size can be determined which bacteria are involved. For example, an E. coli bacteria will grow with big red colonies, and Enterobacter sp. will grow with large dark blue / purple colonies. The sample is seeded with a 10 uL inoculation needle, the lid is applied and the agar plate incubated with the lid down at 35 0C overnight. The plate is read the next day
  Arms: Culture

SUMMARY:
The purpose of this study is to determine whether point-of-care susceptibility testing improve correct choice of antibiotics, clinical and microbiological outcome in patients with uncomplicated urinary tract infection in general practice compared to point-of-care urine culture.

DETAILED DESCRIPTION:
700-900 patients with symptoms of uncomplicated urinary tract infection, consecutively contacting their GP, randomized to either point of care test (POCT) urine culture and empirical treatment or POCT urine culture and susceptibility testing and targeted treatment. Patients are included until 440 with verified positive cultures are included. The two groups are compared with regard to correct choice of antibiotics, clinical remission and microbiological cure rates.

ELIGIBILITY:
Inclusion Criteria:

* Female adult patients
* 18 years or older
* Presenting at their GP with dysuria
* Frequency or urgency, which have been present for 7 days or less and where the GP suspects uncomplicated UTI.
* Patients should be able to deliver a mid-stream urine sample, to provide informed consent and be willing and able to fill out a symptom diary.

Exclusion Criteria:

* Negative dipstick analysis
* Complicated urinary tract infection
* Known pregnancy
* Severe systemic symptoms, high fever, flank pain
* Recent bladder surgery (within past 4 weeks)
* Urinary tract abnormalities
* Serious systemic disease
* Life-threatening cancer
* Insulin dependent diabetes
* Long-term corticosteroid treatment
* Other conditions with compromised immunity
* Former participation in the study
* Patients presenting on a Friday (since the POCT must be read after 24 hours)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The proportion of patients receiving correct treatment | 12 months
  Correct treatment defined as:
  1. If an antibiotic is given, there is significant growth of one or more organisms in the gold standard, which all are sensitive to the given antibiotic. The antibiotic must be one of the recommended first-choice treatments unless the organism(s) is/are resistant to or the patient is allergic
  2. If no antibiotic is given, there is no significant growth in the gold standard

SECONDARY OUTCOMES:
The proportion of patients who are asymptomatic the 4'th day of treatment (clinical cure) | 14 months
-The proportion of patients with no significant bacteriuria on day 14 (bacteriological cure) | 14 months
Accuracy of point-of-care urine culture and susceptibility testing | 14 months
  Accuracy of the two test

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holm, Principal Investigator — Section of General Practice, Dept. of Public Health, University of Copenhagen
Locations (1):
- 21 General practices in Copenhagen area, Copenhagen, Denmark

REFERENCES:
- [Derived] Holm A, Cordoba G, Moller Sorensen T, Rem Jessen L, Frimodt-Moller N, Siersma V, Bjerrum L. Effect of point-of-care susceptibility testing in general practice on appropriate prescription of antibiotics for patients with uncomplicated urinary tract infection: a diagnostic randomised controlled trial. BMJ Open. 2017 Oct 16;7(10):e018028. doi: 10.1136/bmjopen-2017-018028. PMID 29042390
- [Derived] Holm A, Cordoba G, Sorensen TM, Jessen LR, Frimodt-Moller N, Siersma V, Bjerrum L. Clinical accuracy of point-of-care urine culture in general practice. Scand J Prim Health Care. 2017 Jun;35(2):170-177. doi: 10.1080/02813432.2017.1333304. Epub 2017 Jun 1. PMID 28569603
- [Derived] Holm A, Cordoba G, Sorensen TM, Jessen LR, Siersma V, Bjerrum L. Point of care susceptibility testing in primary care - does it lead to a more appropriate prescription of antibiotics in patients with uncomplicated urinary tract infections? Protocol for a randomized controlled trial. BMC Fam Pract. 2015 Aug 21;16:106. doi: 10.1186/s12875-015-0322-x. PMID 26292908